CLINICAL TRIAL: NCT05213754
Title: Acute Ischemic Stroke Registry for Endovascular Treatment in China
Brief Title: Acute Ischemic Stroke Registry for Endovascular Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: AIS-EVT
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Endovascular treatment; Outcome; Registry
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular Treatment — Re-open the occluded cerebral artery using endovascular treatment

SUMMARY:
The Acute Ischemic Stroke Registry for Endovascular Treatment (AIS-EVT) is an academic, prospective, multicenter, observational registry study. Consecutive stroke patients treated with endovascular treatment will be enrolled in stroke centers. Baseline information and clinical follow-up information at 90 days of stroke onset are collected. Data collected include demographics, comorbidities, pathogenesis, blood pressures, stroke severity on admission, time intervals, reperfusion condition, and functional outcome, et al.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute ischemic stroke;
2. Imaging confirmed intracranial large vessel occlusion: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA V4), and posterior cerebral artery (PCA P1);
3. Initiation of any type of endovascular treatment, including intra-arterial thrombolysis, mechanical thrombectomy, aspiration, angioplasty, and stenting;
4. Verbal and written informed consent was provided at the time of admission by patients or their legal authorized representatives.

Exclusion Criteria:

No evidence of large vessel occlusion on digital subtraction angiography.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute ischemic stroke patients with large vessel occlusion receiving endovascular treatment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score at 90 days | 90 days
  The range of the modified Rankin Scale is from 0 to 6. A higher score indicates a worse outcome.
  0-No symptoms; 1-No significant disability; 2-Slight disability; 3-Moderate disability; 4-Moderately severe disability; 5-Severe disability; 6-Dead.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China